CLINICAL TRIAL: NCT05676632
Title: The Impact of Achilles Tendon Rupture on the Structure and Function of the Achilles Tendon and Plantarflexors: a Cross Sectional Analysis
Brief Title: Impact of Achilles Tendon Ruptures: Cross-Sectional Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0882
Record Dates: First submitted 2022-11-10; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-11

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Routine Clinical Care — All participants attending the Achilles Tendon Rupture clinic will receive usual clinical care

SUMMARY:
This project will assess the clinical outcomes of individuals completing rehabilitation for their Achilles tendon rupture at the University Hospitals of Leicester. Patients attending the Achilles tendon rupture clinic or rehabilitation classes will be asked to complete ultrasound imaging, strength testing and questionnaires. This will provide an insight into the rehabilitation outcomes of a broad range of patients at each rehabilitation timepoint.

DETAILED DESCRIPTION:
This study will measure the recovery of participants following Achilles tendon rupture. Measurements will capture individual participants at each rehabilitation time point following Achilles tendon rupture. These time points include following rupture (week 0), after 8 weeks, 10 weeks, 4 months, 6 months and 1 year. The measurements include an ultrasound tissue characterisation scan, isometric (static) strength test and heel raise test. In addition questionnaires will be completed by participants at each time point. Questionnaires include the Achilles Tendon Rupture Score, Hospital Anxiety and Depression Scale, EQ5D (a health related quality of life measure), International Physical Activity Questionnaire, Tampa Scale for Kinesiophobia and the Pain Catastrophising Scale.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* 16 years of age or above

Exclusion Criteria:

* Inability to provide informed consent due to cognitive impairment
* Inability to provide informed consent as unable to understand sufficient English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals attending the Achilles tendon rupture clinic following Achilles tendon rupture
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Tissue Characterisation | Week 0
  Imaging of the Achilles Tendon
Ultrasound Tissue Characterisation | week 8
  Imaging of the Achilles Tendon
Ultrasound Tissue Characterisation | week 10
  Imaging of the Achilles Tendon
Ultrasound Tissue Characterisation | 4 months
  Imaging of the Achilles Tendon
Ultrasound Tissue Characterisation | 6 months
  Imaging of the Achilles Tendon
Ultrasound Tissue Characterisation | 12 months
  Imaging of the Achilles Tendon

SECONDARY OUTCOMES:
Isometric plantarflexor strength testing | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  Isometric plantarflexor strength will be tested in plantargrade (neutral position) using the fysiometer.
Heel Raise Test | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  The heel raise test will measure the amount of heel raises and the work completed by the participant in joules.
Achilles Tendon Rupture Score (ATRS) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  Scores are between 0-100 with a higher score indicating less severe limitations
EuroQol- 5 Dimension - 5 Level (EQ-5D-5L) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  An index score is produced which is calculated using the UK index score reference. The thermometer score is between 0-100 with a higher score indicating better perceived health
Tampa Scale of Kinesiophobia (TSK) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia
Hospital Anxiety and Depression Scale (HADS) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  The two domains (anxiety and depression) provide scores between 0-21 with a higher score indicating higher severity
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or MET minutes representing the amount of energy expended carrying out
Pain Catastrophizing Scale (PCS) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  A total score is calculated from 0-54 with a higher score indicating higher pain catastrophising
36-Item Short Form Survey (SF-36) | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  SF-36 measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). Higher scores indicate higher quality of life
Accelerometer | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  GENEactiv wrist based accelerometer measuring total steps, activity intensity. 24 hours data capture for 7 days
Accelerometer | Week 0, week 8, week 10, 4 months, 6 months and 12 months
  GENEactiv wrist based accelerometer measuring sleep duration for 7 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Briggs-Price S, Yates T, Mangwani J, Bhatia M, Jones A, Mielcarek K, Solaini A, Leung SY, Gravare Silbernagel K, Hebert-Losier K, de Vos RJ, Millar NL, Vicenzino B, O'Neill S. Structure and function of the Achilles tendon and plantarflexors after non-surgical management of Achilles tendon rupture: A cross-sectional study. Musculoskelet Sci Pract. 2026 Feb;81:103459. doi: 10.1016/j.msksp.2025.103459. Epub 2025 Nov 25. PMID 41313926